CLINICAL TRIAL: NCT03677739
Title: Facebook Intervention for Young Onset Melanoma Patients and Families
Brief Title: Young Melanoma Family Facebook Intervention or Healthy Lifestyle Facebook Intervention in Improving Skin Examination in Participants With Melanoma and Their Families
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Sharon Manne, PhD, Professor of Medicine, Rutgers Cancer Institute of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro2018001697; NCI-2018-01741 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Pro2018001697; 131812 (Other: Rutgers Cancer Institute of New Jersey); 1R01CA221854-01A1 (NIH)
Record Dates: First submitted 2018-08-24; First posted 2018-09-19 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Clinical Stage 0 Cutaneous Melanoma AJCC v8; Clinical Stage I Cutaneous Melanoma AJCC v8; Clinical Stage IA Cutaneous Melanoma AJCC v8; Clinical Stage IB Cutaneous Melanoma AJCC v8; Clinical Stage II Cutaneous Melanoma AJCC v8; Clinical Stage IIA Cutaneous Melanoma AJCC v8; Clinical Stage IIB Cutaneous Melanoma AJCC v8; Clinical Stage IIC Cutaneous Melanoma AJCC v8; Clinical Stage III Cutaneous Melanoma AJCC v8; First Degree Relative; Pathologic Stage 0 Cutaneous Melanoma AJCC v8; Pathologic Stage I Cutaneous Melanoma AJCC v8; Pathologic Stage IA Cutaneous Melanoma AJCC v8; Pathologic Stage IB Cutaneous Melanoma AJCC v8; Pathologic Stage II Cutaneous Melanoma AJCC v8; Pathologic Stage IIA Cutaneous Melanoma AJCC v8; Pathologic Stage IIB Cutaneous Melanoma AJCC v8; Pathologic Stage IIC Cutaneous Melanoma AJCC v8; Pathologic Stage III Cutaneous Melanoma AJCC v8; Pathologic Stage IIIA Cutaneous Melanoma AJCC v8; Pathologic Stage IIIB Cutaneous Melanoma AJCC v8; Pathologic Stage IIIC Cutaneous Melanoma AJCC v8

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 Young melanoma Family Facebook focusing on skin cancer (Experimental): Participants join a secret Young melanoma Family Facebook Group and view post messages focusing on skin cancer for 12 weeks.
  Interventions: Other: Informational Intervention; Other: Survey Administration
- Arm 2 Healthy Lifestyle Facebook focusing on healthy lifestyle (Experimental): Participants join a secret Healthy Lifestyle Facebook Group and view post messages focusing on healthy lifestyle for 12 weeks.
  Interventions: Other: Informational Intervention; Other: Survey Administration

INTERVENTIONS:
Other: Informational Intervention — Receive information focusing on skin cancer
  Arms: Arm 1 Young melanoma Family Facebook focusing on skin cancer
Other: Informational Intervention — Receive information on healthy lifestyle
  Arms: Arm 2 Healthy Lifestyle Facebook focusing on healthy lifestyle
Other: Survey Administration — Ancillary studies

SUMMARY:
This trial studies how well Young Melanoma Family Facebook intervention or Healthy Lifestyle Facebook intervention works in improving skin examination in participants with melanoma and their families. Young Melanoma Family Facebook intervention or Healthy Lifestyle Facebook intervention may help improve total cutaneous examinations, skin self-examinations, and sun protection among first degree relatives of young onset participants and the participants themselves.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To examine the efficacy of the Young Melanoma Family Facebook intervention versus the Healthy Lifestyle Facebook intervention on total cutaneous exam (primary outcome), skin self-exam frequency and comprehensiveness, and sun protection practices (secondary outcomes) of first degree relatives (FDRs) of young melanoma survivors.

SECONDARY OBJECTIVES:

I. To examine the efficacy of the Young Melanoma Family Facebook intervention on patients? skin self-exam frequency and comprehensiveness and sun protection habits.

II. To examine the mechanisms of intervention efficacy.

OUTLINE:

PHASE I: Researchers refine content for the Facebook intervention condition and conduct usability testing.

PHASE II: Participants are randomized to 1 of 2 arms.

ARM I: Participants join a secret Young Melanoma Family Facebook Group and view post messages focusing on skin cancer for 12 weeks.

ARM II: Participants join a secret Healthy Lifestyle Facebook Group and view post messages focusing on healthy lifestyle for 12 weeks.

PHASE III: Dissemination planning.

After completion of study, participants are followed up at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* PATIENT: Diagnosed with stage 0-3 melanoma in the last 5 years
* PATIENT: Age at diagnosis 18-39 years
* PATIENT: Completed treatment at least 3 months previously
* PATIENT: Recruited from New Jersey or California State Cancer Registry or MD Anderson Cancer Center
* PATIENT: Does not have a concurrent cancer diagnosis
* PATIENT: Able to speak and read English
* PATIENT: Access to computer, internet, and has a Facebook account
* PATIENT: At least one family member consents
* FDR: Current age 18-80 years
* FDR: Does not have a personal history of melanoma
* FDR: Able to speak and read English
* FDR: Access to computer, internet, and has a Facebook account
* FDR: Has only one FDR with melanoma (patient)
* FDR: Has not had a total cutaneous examination (TCE) in the past 3 years, has done skin self-exam (SSE) fewer than three times in the past year, OR has a sun protection habits average score less than or equal to 4 (?often?)
* FDR: Patient consents

Exclusion Criteria:

* Physical Activity Readiness Questionnaire (Thomas, et. al., 1992): This 7-item scale will be used to screen out individuals who will need to consult a physician for medical clearance before engaging in physical activity. If a participant checks off any of the items, the investigators will ask for a physician clearance before consenting to study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1160 (Estimated)
Dates: Start 2019-06-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Total cutaneous examination (TCE) | At 6 months
  Will be assessed as a binary response (yes/no) did participant have one

SECONDARY OUTCOMES:
Skin Self-exam (Relatives) | Up to 5 years
  Skin self-exam of first degree relatives will be analyzed as a binary (yes/no) Response did participant complete one Yes/No
Skin self-exam - Count Response (Relatives) | Up to 5 years
  Skin self exam of first degree relatives count response will be calculated as frequency/month. Frequency per month reported as a number.
Skin self-exam - Comprehensiveness (Relatives) | Up to 5 years
  : Skin self-exam of first degree relatives comprehensiveness calculated as total # body parts examined during the skin self-exam
Sun Protection Habits (Relatives) | Up to 5 years
  sun protection habits score of first degree relatives will be calculated as continuous variables using the Sun protection behaviors scale (Glanz, et. al., 2002) which measures 5 behaviors (regular outdoor use of: sunscreen, hat, shade, long-sleeved shirt, sunglasses).
Skin self-exam - Count Response (Patients) | Up to 5 years
  Skin self-exam of patients count response calculated as (frequency/month). Frequency per month reported as a number
Skin self-exam - Comprehensiveness (Patients) | Up to 5 years
  Skin self-exam of patients comprehensiveness calculated as total # body parts examined during the skin self-exam.
Sun Protection Habits (Patients) | Up to 5 years
  sun protection habits score of patients will be calculated as continuous variables using the Sun protection behaviors scale (Glanz, et. al., 2002) which measures 5 behaviors (regular outdoor use of: sunscreen, hat, shade, long-sleeved shirt, sunglasses).

OTHER OUTCOMES:
Mediator analyses - Intervention Group | 6 months
  Mediator analyses examining normative influences on the effects of intervention group on TCE, SSE and sun protection.
Mediator analyses - (Relatives) | 6 months
  Mediator analyses examining family and peer support and discussion on the effects of intervention group on TCE, SSE and sun protection.
Mediator analyses - Intervention Group - Risks | 6 months
  Mediator analyses examining risk on the effects of intervention group on TCE, SSE and sun protection.
Mediator analyses - Intervention Group - Benefits | 6 months
  Mediator analyses examining benefits on the effects of intervention group on TCE, SSE and sun protection.
Mediator analyses - Intervention Group - Barriers | 6 months
  Mediator analyses examining barriers on the effects of intervention group on TCE, SSE and sun protection.
Mediator analyses - Intervention Group - Self-efficacy | 6 months
  Mediator analyses examining self-efficacy on the effects of intervention group on TCE, SSE and sun protection.
Mediator analyses - Intervention Group - Change Strategies | 6 months
  Mediator analyses examining use of change strategies on the effects of intervention group on TCE, SSE and sun protection.
Moderator analysis - Melanoma Risk Factors | 6 months
  Moderator analysis Melanoma risk factors will explore whether the intervention group is more effective for subsets of FDRs.
Moderator analysis - month of the year enrolled | 6 months
  Moderator analysis month of the year enrolled will explore whether the intervention group is more effective for subsets of FDRs.
Moderator analysis - Residential Latitude | 6 months
  Moderator analysis residential latitude will explore whether the intervention group is more effective for subsets of FDRs.
Moderator analysis - Sex | 6 months
  Moderator analysis sex will explore whether the intervention group is more effective for subsets of FDRs.
Moderator analysis - patient disease stage | 6 months
  Moderator analysis patient disease stage will explore whether the intervention group is more effective for subsets of FDRs.
Moderator analysis relationship to patient | 6 months
  Moderator analysis relationship to patient will explore whether the intervention group is more effective for subsets of FDRs.
Predictor - Engagement | 6 months
  Facebook engagement including likes, comments- collected at the end of the group
Predictor - Social Network Use | 6 months
  Social network use measured by self-reported frequency of use of popular social media sites

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Manne, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (2):
- United States (2):
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Manne S, Pagoto S, Peterson S, Heckman C, Kashy D, Berger A, Studts C, Negron R, Buller D, Paddock L, Gallo J, Kulik A, Frederick S, Pesanelli M, Domider M, Grosso M. Facebook Intervention for Young-Onset Melanoma Survivors and Families: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2023 Jan 24;12:e39640. doi: 10.2196/39640. PMID 36692933

DOCUMENTS (1):
  • Informed Consent Form (2024-09-16): https://cdn.clinicaltrials.gov/large-docs/39/NCT03677739/ICF_000.pdf